CLINICAL TRIAL: NCT02539472
Title: Evaluation of a Combination of Blood Biomarkers for the Early Diagnosis of Mycosis Fungoides
Brief Title: Early Diagnosis of Mycosis Fungoides
Acronym: DIAPREMYF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K14097
Record Dates: First submitted 2015-07-20; First posted 2015-09-03 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- investigation (Experimental): Blood sampling for quantitative evaluation of nine candidate biomarkers (CD158k/KIR3DL2, KIR2DL4, KIR2DS1, KIR2DS3, KIR3DL1, NKp46, PLS3/T-Plastin, Twist and TOX) by quantitative RT-PCR.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling for quantitative evaluation of nine candidate biomarkers (CD158k/KIR3DL2, KIR2DL4, KIR2DS1, KIR2DS3, KIR3DL1, NKp46, PLS3/T-Plastin, Twist and TOX) by quantitative RT-PCR.

SUMMARY:
Mycosis fungoides (MF) is an epidermotropic cutaneous T cell lymphoma characterized by the accumulation of CD4+ T-lymphocytes in the skin. Early MF presents as erythematous patches and/or infiltrated plaques. The diagnosis of early MF is a major diagnostic challenge and the differential diagnosis with inflammatory dermatoses is often very difficult. The histopathological diagnosis is also difficult and delayed. Therefore, it is important to develop biomarkers and/or a combination of biomarkers in order to improve the early diagnostic of MF.

In a previous trial, investigators included 490 patients in a study aiming at identifying skin biomarkers of early MF. Several activating and inhibiting KIRs were found to be interesting for the skin diagnostic of MF, mainly KIR2DL4 and KIR3DL2. Investigators later evaluated blood biomarkers in patients with erythrodermic MF and Sezary Syndrome (SS). This French institutional study demonstrated that the identification by PCR of a combination of 4 blood markers (CD158k/KIR3DL2, PLS3/T-Plastin, Twist and NKp46) allowed a reliable diagnosis of lymphoma in erythrodermic patients. This previously published study interestingly showed that 30% to 50% of patients with early MF expressed at least one of these biomarkers in the blood (unpublished data). Other groups also recently showed that TOX can be a diagnostic tool for MF.

The aim of this study is to establishing an accurate blood diagnosis for early suspected MF by demonstrating that newly identified biomarkers or their combination [5 cutaneous KIR receptor markers (KIR2DS1, KIR2DS3, KIR3DL1, KIR2DL4, KIR3DL2) and 5 blood biomarkers (TOX, Twist-1, PLS3/T-plastin, KIR3DL2, NKp46)] are differentially expressed by patients with MF and patients with inflammatory dermatoses closely resembling MF lesions.

Statistical analysis will establish the best combination of blood biomarkers allowing the differentiation between the two groups of patients, combination that could represent a suitable diagnostic tool for early MF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with erythematous dermatitis of subacute evolution (> 15 d) or chronic evolution, in the form of patches/plaques, leading to a clinically suspected cutaneous T cell lymphoma
* Free and informed consent signed
* Erythematous dermatosis, sub-acute (> 15 days) or chronic, suspicious of MF
* Lack of previous hemopathy or cutaneous or extra-cutaneous lymphoma
* Age > 18 years
* A skin biopsy for routine diagnostic histopathological analysis at the time of inclusion
* With an analysis of T-cell clonality in blood and skin at the time of inclusion

Exclusion Criteria:

* Children under 18 years
* Sick adults under guardianship
* Patients refusing to participate in the research protocol
* Subjects not affiliated with the national health insurance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Early MF Benign inflammatory dermatoses | 12 months

SECONDARY OUTCOMES:
Percentage of positivity of each marker | 12 months
  [5 cutaneous KIR receptor markers (KIR2DS1, KIR2DS3, KIR3DL1, KIR2DL4, KIR3DL2) and 5 blood biomarkers (TOX, Twist-1, PLS3/T-plastin, KIR3DL2, NKp46)]

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, Paris, France